CLINICAL TRIAL: NCT03692702
Title: Wellness Enhancing Physical Activity for Young Children Preschool Teacher Training
Brief Title: Wellness Enhancing Physical Activity for Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Jessica Hoffman, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WEPLAY
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WE PLAY (Experimental): Teachers in this condition received the WE PLAY training.
  Interventions: Behavioral: WE PLAY
- Control (No Intervention): Preschools in this condition received the same physical activity equipment that preschools in the WE PLAY condition received. Teachers were not provided with any specific instructions or information about physical activity.

INTERVENTIONS:
Behavioral: WE PLAY — WE PLAY is an online preschool teacher training that is based in theory and implementation science. It contains six components: (1) online training; (2) video library; (3) game sheets; (4) teacher self-assessment; (5) supervisor support; and (6) activity packs containing low cost physical activity equipment
  Arms: WE PLAY

SUMMARY:
Wellness Enhancing Physical Activity for Young Children (WE PLAY) is a teacher training that is based online and was designed to support early childhood educators' efforts to promote physical activity (PA) through structured and unstructured active play with preschoolers. WE PLAY includes six components: (1) online training; (2) video library; (3) game sheets; (4) teacher self-assessment; (5) supervisor support; and (6) activity packs that are designed to work synergistically. The purpose of this study was to examine the impact of WE PLAY on children's levels of moderate to vigorous physical activity (MVPA) during school hours. We hypothesized that children whose teachers received WE PLAY would have higher levels of MVPA during school hours at post-intervention relative to pre-intervention and relative to children whose teachers did not receive WE PLAY. A second purpose was to examine the impact of WE PLAY on teacher outcomes (i.e., knowledge, intentions, perceived behavior control, subjective norms, perceived power beliefs, normative beliefs, and moral norms). We hypothesized that teachers who participated in WE PLAY would demonstrate higher scores on each of these variables at post-intervention relative to pre-intervention and to teachers in the control group. A cluster randomized controlled trial was used in this study. Six Head Start preschools were pair matched and randomized to the intervention (WE PLAY) or control groups. Preschool children (N=57) and their teachers (N=25) participated. Child MVPA was measured using accelerometers for 5-day periods at pre- and post-intervention. Teacher variables were measured using online surveys.

ELIGIBILITY:
Inclusion Criteria:

* All teachers at the participating programs, and all children within the participating teachers' classrooms, were eligible to participate in this study.

Exclusion Criteria:

* There were no exclusion criteria based on gender, race/ethnicity, language spoken at home, socio-economic level, or any other demographic variable.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) per minute in children | Pre-intervention was in week 1 and post-intervention was in week 4
  We measured child PA using ActiGraph GT9X Link monitors for 24-hour periods across five days at both pre-intervention and post-intervention

SECONDARY OUTCOMES:
Change in teacher knowledge | Pre-intervention (week 1; both groups). The WE PLAY group's knowledge was assessed again immediately following the online training (week 2). The control group's knowledge was measured a second time at the post-intervention assessment (week 4).
  12 knowledge items were developed for this study and were drawn from content covered in the online training. Scores ranged from 0-12. Higher scores indicate higher levels of knowledge.
Change in perceived behavioral control | Pre-intervention (week 1) and post-intervention (week 4)
  Items (n=4) were from a previously developed scale. Scores ranged from 4-24. Higher scores indicate more positive perceptions about one's ability to promote physical activity with students.
Change in subjective norms | Pre-intervention (week 1) and post-intervention (week 4)
  Items (n=3) were from a previously developed scale. Scores ranged from 3-18. Higher scores indicate that promoting physical activity with children is viewed as important by the people most important to the respondent.
Change in moral norms | Pre-intervention (week 1) and post-intervention (week 4)
  Items (n=4) were from a previously developed scale. Scores ranged from 4-24. Higher scores indicate a stronger moral obligation to promote physical activity with students.
Change in normative beliefs | Pre-intervention (week 1) and post-intervention (week 4)
  Items (n=5) were from a previously developed scale. Scores ranged from 5-30. Higher scores indicate that important people surrounding the respondent think that promoting physical activity with students is important.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Hoffman, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States